CLINICAL TRIAL: NCT06685679
Title: Melatonin as an Adjunct Therapy to Milrinone for Pulmonary Hypertension in Full Term Neonates
Brief Title: Melatonin for Pulmonary Hypertension in Full Term Neonates
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Ibrahim, Assistant professor of pediatrics, Ain shams university, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Melatonin in pulmonary hyperte
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2024-11

CONDITIONS: Neonatal Diseases and Abnormalities; Neonatal Mortality; Pulmonary Arterial Hypertension; Pulmonary Arterial Hypertension, Children
Keywords: Neonate; Pulmonary hypertension; Melatonin; Milrinon
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group melatonin group (Experimental): Intervention group : will receive oral melatonin (Kids Daily Vit Sleep syrup) 3 mg/kg/day divided in 3 doses , after enteral feeding, for 3 consecutive days, as combined therapy to milrinone (Garofoli et al., 2021).
  Human studies documented that short-term use of melatonin is safe, even in extreme doses (Andersen et al., 2016).
  Interventions: Drug: Melatonin
- Control group (Placebo Comparator): Control group: will receive the treatment of PHN as our NICU protocol in the form of loading dose of milrinone (50 μg/kg) over 60 mins followed by a maintenance infusion (0.33-0.99 μg/kg/min) for 72 hrs. (McNamara et al., 2013) And equivalent amout of distilled water as a placebogive at same time intervals as melatoni
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Melatonin — oral melatonin 3 mg/kg/day divided in 3 doses , after enteral feeding, for 3 consecutive days, as combined therapy to milrinone
  Arms: Intervention group melatonin group
Other: Placebo — Equivalent amount of distilled water will be given every hours as combined therapy to milrinone
  Arms: Control group

SUMMARY:
Published evidence has provided a possible role of melatonin and the treatment of pulmonary hypertension through its strong antioxidant properties and improving vascular function in animals.

This study will test the hypothesis of the possible use of melatonin as an adjunct therapy to milrinone for neonatal pulmonary hypertension.

DETAILED DESCRIPTION:
Normal pulmonary artery pressure shows a gradual declining trend after birth, and pulmonary artery pressure of 72 h after birth is still higher than that of normal adults Infants born after 34 weeks of gestation with primary findings on physical examination reveals tachypnoea, retractions, grunting, desaturation unresponsive to supplemental O2, cyanosis and pulmonary arterial pressure (PAP) > 25 mm Hg measured by echocardiography, within 72 h of birth, are considered to have pulmonary hypertension Pulmonary hypertension in neonates (PPHN) is a syndrome characterized by failure in the mechanisms that decrease pulmonary vascular resistance (PVR) and pulmonary arterial pressure (PAP) after birth Persistent pulmonary hypertension of newborn (PPHN) develops when pulmonary vascular resistance (PVR) remains elevated after birth, resulting in right-to-left shunting of blood through fetal circulatory pathways. The PVR may remain elevated due to pulmonary hypoplasia, like that seen with congenital diaphragmatic hernia, and maladaptation of the pulmonary vascular bed as occurs with perinatal asphyxia It has been shown that one of the mechanisms involved in the pathophysiology of PPHN is oxidative stress, which results in an imbalance between an increase in free radicals generation and decreased antioxidant capacity Currently, the treatment for PHN considers timely and precise interventions such as intravenous milrinone, oral pulmonary vasodilators such as endothelin receptor antagonist, phosphodiesterase-5 inhibitors such as sildenafil, inhaled nitric oxideand are used both during acute and chronic phases of PPHN, controlled oxygen administration, and even extracorporeal membrane oxygenation.

However, these therapeutic strategies do not markedly reduce the mortality and the long-term neonatal outcomes remain poor Melatonin, more commonly known as the sleep hormone, has been highlighted by experimental evidence, to have significant effects as a direct scavenger of oxygen free radicals and induces antioxidant enzymatic It has been shown that melatonin has vasodilator properties and may modulate pro-oxidant sources in the neonatal lung which is proposed to treat PHN in the first days of neonatal life.

ELIGIBILITY:
Inclusion Criteria:

* full term neonates ≥37 weeks diagnosed with pulmonary hypertension, with Pulmonary arterial pressure (PAP) > 25 mm Hg measured by echocardiography, within 72 h of birth (Chetan et al., 2022).

Exclusion Criteria:

* Neonates with major congenital anomalies like congenital heart diseases

  * NPO or any contraindications to oral intake
  * Neonates with suspected inborn error of metabolism

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Pulmonary arterial pressure | After 72 hours of the start of the drug
  Measuring pulmonary artery pressure by echocardiography
FiO2 | Hourly for 3 days
  FiO2 needs to maintain oxygen saturation monitored non invasively

SECONDARY OUTCOMES:
Hospital stay | One month
  Duration of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Information can be shared upon accepted request

REFERENCES:
- [Background] Chetan C, Suryawanshi P, Patnaik S, Soni NB, Rath C, Pareek P, Gupta B, Garegrat R, Verma A, Singh Y. Oral versus intravenous sildenafil for pulmonary hypertension in neonates: a randomized trial. BMC Pediatr. 2022 May 27;22(1):311. doi: 10.1186/s12887-022-03366-3. PMID 35624452
- [Background] 1- Andersen LPH., Gögenur I, Rosenberg J, Reiter RJ. The safety of melatonin in humans. Clin Drug Investig. 2016 Mar. 36(3), 169-175. 2- Ballard JL, Khoury JC, Wedig K, Wang L, Eilers-Walsman BL and Lipp R. New Ballard Score, expanded to include extremely premature infants. J pediatr. 1991 sep. 119(3), 417-423. 3- Chetan C, Suryawanshi P, Patnaik S, Soni NB, Rath C, Pareek P,et al. Oral versus intravenous sildenafil for pulmonary hypertension in neonates: a randomized trial. BMC pediatr . 2022 May . 22(1), 1-7. 4- D'Angelo, G., Chimenz, R., Reiter, R. J., & Gitto, E. Use of melatonin in oxidative stress related neonatal diseases. Antioxidants. 2020, 9(6), 477